CLINICAL TRIAL: NCT01255319
Title: Conditioning With Cyclophosphamide, Fludarabine and Antithymocyte Globulin for Allogeneic Hematopoietic Cell Transplantation in Lower Risk Myelodysplastic Syndrome
Brief Title: Cyclophosphamide, Fludarabine and Antithymocyte Globulin Conditioning in Myelodysplastic Syndrome (MDS)
Acronym: CyFluATG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Other Study IDs: Allo-038
Record Dates: First submitted 2010-11-30; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the feasibility and efficacy of the conditioning regimen with cyclophosphamide, fludarabine and antithymocyte globulin (CyFluATG) for allogeneic hematopoietic cell transplantation (HCT) in patients with lower risk myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
Conditioning therapy

* Cytoxan 50 mg/kg/d on d-3 to -2
* Fludarabine 30 mg/m2 on d-6 to -2
* Antithymocyte globulin (ATG; Thymoglobulin®) 1.5 mg/kg/d (for HLA-matched sibling donor HCT) or 3.0 mg/kg/d (for other alternative donor HCT)
* Methylpd 2 mg/kg/d on d-4 to -1

Mobilization and harvest

* G-CSF 10 mcg/kg/d s.c. on d-3 to 0
* Harvest of PBMCs on d 0 to +1

Donor G PBMC infusion

* Infuse G-PBMCs on d 0 to d+1.

GVHD prophylaxis

* Cyclosporine 1.5 mg/kg i.v. q 12 hrs beginning on d-1 and changed to oral dosing (with twice the i.v. dose) when oral intake is possible. Tapered beginning between d+30 and d+60.
* Methotrexate 15 mg/m2 i.v. on d+2, and 10 mg/m2 i.v. on d+4 and d+7

Preemptive dose-escalating DLIs

* Begin at d+120 or at least 2 wks after IST discontinuation.
* Failure to achieve full donor chimerism No evidence of GVHD
* CD3+ cell dose increment q 4 wks -+ cell dose: HLA-matched donor HCT (1 x 107/kg, 5 x 107/kg, 1 x 108/kg), HLA-matched unrelated donor HCT (1 x 106/kg, 5 x 106/kg, 1 x 107/kg), HLA-matched familial donor HCT (1 x 105/kg, 5 x 105/kg, 1 x 106/kg)

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower risk MDS (bone marrow blast percentage < 5%)
* Patients with appropriate hematopoietic cell donor
* Adequate performance status (Karnofsky score of 70 or more; see Appendix II)
* Adequate hepatic and renal function (AST, ALT, and bilirubin < 3.0 x upper normal limit, and creatinine < 2.0 mg/dL).
* Adequate cardiac function (left ventricular ejection fraction of 40% or more on heart scan or echocardiogram)
* Signed and dated informed consent must be obtained from both recipient and donor.

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lower risk MDS
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
feasibility and efficacy | 4years
  To evaluate the feasibility and efficacy of the conditioning regimen with cyclophosphamide, fludarabine and antithymocyte globulin (CyFluATG) for allogeneic hematopoietic cell transplantation (HCT) in patients with lower risk myelodysplastic syndrome (MDS). The efficacy of the treatment will be measured in terms of engraftment and non-relapse mortality (the primary endpoints)

SECONDARY OUTCOMES:
progression-free survival, and overall survival | 4 years
  This study will also evaluate donor chimerism, secondary graft failure, acute and chronic graft-versus-host disease (GVHD), immune recovery, infections, progression-free survival, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Je-Hwan Lee, Doctor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Asanbyeongwon-gil, Songpa-gu, South Korea

REFERENCES:
- See also: Conditioning with cyclophosphamide, fludarabine and antithymocyte globulin for allogeneic hematopoietic cell transplantation in lower risk myelodysplastic syndrome — http://www.google.co.kr